CLINICAL TRIAL: NCT06920979
Title: Stop Sepsis Through Home Monitoring Cooperative
Acronym: Stethoscoop
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Guy Hans, Clinical Professor, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EDGE003963; Governement Health Belgium (Other: Stethoscoop federal governement heatlh Belgium)
Record Dates: First submitted 2025-03-19; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Home Monitoring Follow-up; Infection; Innovativeness
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- (semi)continue monitoring of patients at risk for sepsis at home (Other): Patients with acute infections at risk of developing sespsis will be followed in their home setting using wearables that provide (semi-)continue monitoring of vital signs as well as through follow up using a desingated smarthphone application.
  Interventions: Other: (semi)continue monitoring of patients at risk for sepsis at home

INTERVENTIONS:
Other: (semi)continue monitoring of patients at risk for sepsis at home — (semi)continue monitoring of patients at risk for sepsis at home

SUMMARY:
In this study, patients presenting with acute infections at risk of developing sepsis will be followed in their home setting using wearables that provide (semi-)continue monitoring of vital signs as well as through follow up using a designated smartphone application. This is an innovative pilot study that will examine the potential of transmural care through telemonitoring for the first time in patients at risk for developing sepsis. By allowing for active follow-up of vital parameters in a transmural setting, this project aims to reduce the number of hospitalizations as compared to current practice. Furthermore, we aim to the number of patients referred to the emergency department after a visit at their primary care physician. Thereby, we aim to reduce the healthcare burden, yet providing the ability for rapid intervention in case of detarioration of patients, thereby reducing morbidity and mortality as well as associated costs.

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients aged 18 years or older, capable of giving informed consent, presenting with signs of severe acute infection with a risk of developing sepsis at the emergency department or at their primary care physician.

Exclusion Criteria:

* Patients that are severely ill and require immediate hospitalization Qucik Sepsis Related Organ Failure score (QSOFA) ≥ 1 National Early Warning Score (NEWS) ≥ 5
* Patients that demonstrate confusion, changes in mental state and/or an Mini-Mental State Examination (MMSE) below 26
* Presence of neuropenic fever
* Patients currently undergoing immunosuppressive therapy or chemotherapy
* Patients with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS)
* Suspicion of appendicitis, suspicion of meningitis or meningeal irritation, suspicion of or high risk of developing endocarditis
* Complicated operation wounds at the time of screening
* Proven pneumonia (CURB 65 score ≥ 1)
* Emphysema, Chronic Obstructive Pulmonary Disease (COPD) GOLD >1 or interstitial lung disease
* Patients with oxygen at home > 2 l/min on a chronic basis (severe underlying lung disease?)
* Severe cardiovascular disease including:

  * Severe heart failure New York Heart Association (NYHA) class > 1
  * Endoprosthesis
  * Cardiac arrhythmia including atrial fibrillation
  * Severe heart valve abnormalities
  * Mechanic valve replacement
  * Recent acute myocardial infarct or coronarography (less than 1y ago)
  * Severe peripheral vascular morbidity
* Acute chest pain (suspicion of acute coronary pathology)
* Suspicion of/chance of septic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the development and roll out of a central medical center for monitoring at home | From enrollment to the end of monitoring depending on the clinical evolution of the patient, with a minimum of one week and a maximum follow-up of three weeks.
  The total number of patients who use the home monitoring system for at least three days. This measure evaluates the adoption and feasibility of remote monitoring within a real-world setting.
Evaluation of the development and roll out of a central medical center for monitoring at home | From enrollment to the end of monitoring depending on the clinical evolution of the patient with a minimum follow-up of one week and up to a maximum of three weeks.
  The proportion of patients whose wearable devices and smartphone applications successfully capture at least 80% of the required physiological data over the home monitoring period. This assesses the reliability and consistency of the telemonitoring system.
Evaluation of the development and roll out of a central medical center for monitoring at home | From enrollment to the end of monitoring depending on the clinical evolution of the patient with a minimum follow-up of one week and up to a maximum of three weeks of follow-up.
  The effectiveness of telemonitoring wearables and smartphone applications in accurately measuring and tracking the National Early Warning Score (NEWS) in a home setting. This evaluates the clinical utility of remote patient monitoring for early detection of health deterioration.
Evaluation of the development and roll out of a central medical center for monitoring at home | From enrollment to the end of monitoring depending on the clinical evolution of the patient with a minimum follow-up of one week and up to a maximum of three weeks of follow-up.
  The number of emergency departments and primary care physicians actively using the telemonitoring platform to access and review patient data. This assesses the level of integration of home monitoring into routine clinical workflows.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital (UZA), Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The results will be published in a research paper in a scientific journal.